CLINICAL TRIAL: NCT03775447
Title: FoxBioNet: ECV (Extracellular Vesicle) 003
Brief Title: Fox BioNet Project: ECV-003
Status: Completed | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: University Health Network, Toronto (Other); Indiana University (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Connie Marras, Neurologist at Toronto Western Hospital Movement Disorders Centre, University Health Network, Toronto
Other Study IDs: ECV-003
Record Dates: First submitted 2018-11-20; First posted 2018-12-14 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Biomarker; LRRK2; CSF
MeSH Terms: conditions — Parkinson Disease | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cerebro-Spinal Fluids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Disease Patients: * A diagnosis of Parkinson's disease in the opinion of the enrolling investigator
  * Disease duration: any
  * Male or female age 18 years or older at time of PD diagnosis.
  Interventions: Procedure: Lumbar Puncture
- Healthy Control (HC) Subjects: • Male or female age 18 years or older at Screening.
  Interventions: Procedure: Lumbar Puncture

INTERVENTIONS:
Procedure: Lumbar Puncture — Lumbar Puncture for collection of Cerebrospinal Fluids
  Other Names: Biofluid Samplings: Blood

SUMMARY:
The goal of this study is to optimize pre-analytical cerebrospinal fluid (CSF) extracellular vesicle isolation protocols for increasing the detection of LRRK2 activity in human CSF

DETAILED DESCRIPTION:
Specific aims to accomplish this objective are:

PRIMARY OBJECTIVES:

* To evaluate a series of extracellular vesicle isolation methods for their ability to enrich for LRRK2 and increase the detection of LRRK2 in CSF samples.
* To compare the measurements of LRRK2, p1292 LRRK2, Rabs and pRabs from the ECVs isolated using each method.
* To assess the inter-lab reliability of each method

SECONDARY OBJECTIVES

* To assess the ability of the network of sites to efficiently conduct a study involving biosample collection for PD research. Efficiency will be assessed using measures of the time taken to meet specific milestones within the study
* To assess the ability of the network to collect high quality biospecimens adhering to agreed-upon protocols.
* To gauge the willingness of participants to participate in subsequent Fox BioNet studies

ELIGIBILITY:
Inclusion Criteria:

Parkinson's Disease Patients:

* A diagnosis of Parkinson's disease in the opinion of the enrolling investigator
* Disease duration: any
* Male or female age 18 years or older at time of PD diagnosis.

Healthy Controls:

•Male or female age 18 years or older at Screening.

Exclusion Criteria:

Parkinson's Disease Patients:

* Inability to provide informed consent
* Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans.

Healthy Controls:

* Inability to provide informed consent
* Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans.
* Currently pregnant (female participants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 36 subjects will be enrolled to participate in this study, a combination of Parkinson Disease (PD) (any stage) and Healthy Controls in no specified proportion.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
degree of LRRK2 enrichment achieved. The measure will vary depending on the method of LRRK2 enrichment used | 1 year
  For methods involving immunoprecipitation: Increase in peptide spectral matches on mass spectrometry For methods amenable to antibody-based detection: increase in LRRK2 intensity on Western blotting (arbitrary units).

SECONDARY OUTCOMES:
Power analysis to guide future research | 1 year
  Pilot data to enable calculations for power analysis to guide future research studies for the primary outcomes
Time from IRB submission to approval by central IRB | 3 months
  Time from IRB submission to approval by central IRB
Time from central IRB approval to site approval | 3 months
  Time from central IRB approval to site approval (for those sites requiring administrative review)
Time from site selection to contract full execution | 4 months
  Time from site selection to contract full execution
Completion of Recruitment | 6 months
  Time from site activation to completion of recruitment.
Proportion of samples conforming to collection | 6 months
  Proportion of samples conforming to collection, processing and shipping protocols.
Retention | 1 year
  Proportion of participants agreeing to be contacted for future Fox BioNet protocols

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No